CLINICAL TRIAL: NCT04814719
Title: An Observational Follow-up Study to Investigate the Duration of Treatment Effect With Subcutaneous Injections of Pentosan Polysulfate Sodium Compared With Placebo in Adult Participants With Knee Osteoarthritis Pain
Brief Title: Treatment and Duration Effect of Pentosan Polysulfate Sodium (PPS) in Participants With Knee Osteoarthritis Pain
Status: Completed | Type: Observational
Sponsor: Paradigm Biopharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PARA_OA_006
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Pentosan Sulfuric Polyester; Sodium Chloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pentosan Polysulfate Sodium: Pentosan Polysulfate Sodium (PPS) at Dose and frequency selected in Stage 1 of Parent Study for 6 weeks
  Interventions: Drug: Pentosan Polysulphate Sodium
- Placebo: Placebo for 6 weeks
  Interventions: Drug: Placebo (Sodium Chloride Injection, 0.9%)

INTERVENTIONS:
Drug: Pentosan Polysulphate Sodium — Subcutaneous Injection (100mg/ml)
  Other Names: PPS
  Groups: Pentosan Polysulfate Sodium
Drug: Placebo (Sodium Chloride Injection, 0.9%) — Placebo to match PPS
  Other Names: Sodium Chloride
  Groups: Placebo

SUMMARY:
The purpose of this study is to measure the duration of treatment effect with subcutaneous injections of pentosan polysulfate sodium (PPS) compared with placebo in adult participants with knee osteoarthritis (OA) pain. The study duration will be up to 34 weeks.

Participants who completed pDay 162 of Study PARA_OA_002 (i.e. did not discontinue/withdraw prematurely from the parent study) will be invited to participate.

DETAILED DESCRIPTION:
This is an observational study to determine duration of treatment effect and assess long-term safety up to 52 weeks post PPS use for 6 weeks in parent study (PARA_OA_002). The duration of treatment effect will be evaluated by the OMERACT-OARSI responder criteria for knee OA.

Eligible participants will be enrolled in Study PARA_OA_006 at the completion of the parent study PARA_OA_002. There will be no intervention in this observational study.

Participants will attend screening (visit 1), three phone visits at 8, 16, and 24 weeks, and an EOS (end of study) visit 34 weeks at the site, a total of 5 visits. Participants questionnaires include WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) NRS 3.1 Index, PGIC (Patients Global Impression of Change), WPAI (Work Productivity and Activity Impairment) and quality of life SF-36.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed Day 168 of Study PARA_OA_002 (ie, did not discontinue/withdrew prematurely from the parent study).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

• An employee of the Sponsor, clinical research organisations or research site personnel directly affiliated with this study or their immediate family members defined as a spouse, parent, sibling, or child, whether biological or legally adopted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who completed pDay 168 of Study PARA_OA_002 (ie, did not discontinue/withdraw prematurely from the parent study).
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2023-06-24 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Assess duration of treatment effect of PPS in participants with OA pain | From initial response time baseline in parent study up to 34 weeks
  Time from initial response in the parent study (PARA_OA_002) to loss of OMERACT-OARSI (Outcomes Measures in Rheumatology - Osteoarthritis Research Society International) response.

SECONDARY OUTCOMES:
Assess duration of treatment effect of PPS in participants with OA pain | Week 8, 16, 24, and 34
  Percentage of participants considered OMERACT- OARSI (Outcomes Measures in Rheumatology - Osteoarthritis Research Society International) responders at each timepoint..
Assess efficacy of PPS treatment on knee pain in participants with knee OA pain | Baseline (parent study) pDay1, weeks 8, 16, 24, and 34
  WOMAC NRS 3.1 (Western Ontario and McMaster Universities Osteoarthritis Index) Index Pain average subscale score. Reduction in knee pain of ≥30% and ≥50% as assessed by the average pain WOMAC NRS 3.1 subscale score. Ranges 0-10 with 0 represents no pain and 10 represents extreme pain.
WOMAC NRS 3.1 (Western Ontario and McMaster Universities Osteoarthritis Index) assessment of knee function in participants with knee OA pain | Baseline (parent study) pDay1, weeks 8, 16, 24, and 34
  WOMAC NRS 3.1 Index Function WOMAC NRS 3.1 Index.. Improvement of function assessed of ≥30% and ≥50% as assessed by the average Function subscale score (knee) during the past 48 hours. Ranges Scoring 0-10, 0 is better or none and 10 is worse.
WOMAC NRS 3.1 (Western Ontario and McMaster Universities Osteoarthritis Index) knee stiffness assessment in participants with knee OA | Baseline (parent study) pDay1, weeks 8, 16, 24, and 34
  WOMAC NRS 3.1 Index Stiffness average subscale score. Ranges 0-10, 0 is better or none and 10 is extreme or worse.
Overall score WOMAC NRS 3.1 (Western Ontario and McMaster Universities Osteoarthritis Index) in participants with knee OA | Baseline (parent study) pDay1, weeks 8, 16, 24, and 34
  WOMAC NRS 3.1 Index Overall average subscale score The WOMAC® NRS 3.1 Index consists of 24 questions and produces 3 sub-scales scores for pain (5 questions), stiffness (2 questions), and function (17 questions) and a total score that summarizes overall disability. Score of 0 is better and the higher score is worse
Assess effect of PPS on Patient Global Impression of Change (PGIC) in participants with knee OA pain | Weeks 8, 16, 24 and 34
  The PGIC is a self-administered question that rates participants overall improvement in chronic pain since beginning treatment from 1 "no change (or condition has worsened)" to 7 "a great deal better" in response to the question "Since beginning treatment, how would you describe the change (if any) in activity, limitation, symptoms, emotions, and overall QoL related to your arthritis".
Change from baseline of the parent study in Quality of Life (QoL) as assessed by Short Form-36 General Health Survey (SF-36) | Baseline (parent study) pDay1, Weeks 8, 16, 24 and 34
  The SF-36 v2 is a 36-item, patient-reported survey of patient health, consisting of 8 scaled scores, which are the weighted sums of the questions in their section. The 1-week recall form asks the respondent to answer the questions as they pertain to the way he or she felt or acted during the past week. Score ranges 0-100 higher scores indicate better health.
Change from baseline of the parent study in Work Productivity and Activity Impairment (WPAI) questionnaire. | Baseline (parent study) pDay1, Weeks 8, 16, 24 and 34
  This WPAI questionnaire (WPAI:OA-knee) is a validated self-administered questionnaire that assesses work impairment due to OA . The questionnaire gathers information on employment status, hours worked, hours missed due to OA, and hours missed for any other reasons
Assess real-world use of pain medications/therapies, following a single course of PPS | Baseline up to Week 34
  Number of days rescue medication used or use of other pain medications and therapies
Incidence of treatment-emergent AE's, SAE's and AESI of PPS is participants with knee OA pain | Baseline up to Week 34
  Data of SAE's, AE's, causally to IP, AE's of Special Interest (AEST), AE's requiring any intervention for index knee pain and AE's requiring pain medication.

OTHER OUTCOMES:
Change in subchondral Bone Marrow Lesion (BML) on Magnetic Resonance Imaging (MRI) from baseline of the parent study. | Baseline (parent study) pDay1 and at Week 34
  MRIs will be reviewed by an independent trained reader blinded to participant characteristics, study information and timing of MRI scans. All measurement will be done in duplicate
Change in joint synovitis/effusion volume on MRI | Baseline (parent study) pDay1 and at Week 34
  MRIs will be reviewed by an independent trained reader blinded to participant characteristics, study information and timing of MRI scans. All measurement will be done in duplicate
Effect of PPS on Change in cartilage volume on MRI | Baseline (parent study) pDay1 and at Week 34
  MRIs will be reviewed by an independent trained reader blinded to participant characteristics, study information and timing of MRI scans. All measurement will be done in duplicate
Change in bone shape on MRI and whether these correlate with clinical outcomes | Baseline (parent study) pDay1 and at Week 34
  MRIs will be reviewed by an independent trained reader blinded to participant characteristics, study information and timing of MRI scans. All measurement will be done in duplicate
Change in joint space width on X-ray | Baseline (parent study) pDay1 and at Week 34
  X-Rays will be reviewed by an independent trained reader blinded to participant characteristics, study information and timing of MRI scans. All measurement will be done in duplicate
Change in joint space width on MRI | Baseline (parent study) pDay1 and at Week 34
  MRIs will be reviewed by an independent trained reader blinded to participant characteristics, study information and timing of MRI scans. All measurement will be done in duplicate
Explore any correlation between joint space width measurements from x-rays and MRI | Week 34
  MRIs and x-rays will be reviewed by an independent trained reader blinded to participant characteristics, study information and timing of MRI scans and x-rays. All measurement will be done in duplicate.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schnitzer, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (2):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States
- Emeritus Research, Camberwell, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No